CLINICAL TRIAL: NCT07223645
Title: Handgrip Training and Brain Blood Flow Regulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Joseph Watso, Laboratory Director, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00006271
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Inactivity/Low Levels of Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Isometric Handgrip Training - Intervention (Experimental): Participants will perform moderate-intensity handgrip training three days per week for eight weeks using a handheld device.
  Interventions: Device: Handgrip Training
- Isometric Handgrip Training - Sham (Sham Comparator): Participants will perform very low-intensity handgrip training three days per week for eight weeks using a handheld device.
  Interventions: Device: Handgrip Training

INTERVENTIONS:
Device: Handgrip Training — Handgrip training 3 days per week for 8 weeks

SUMMARY:
This study aims to investigate the effect of isometric handgrip training on brain blood vessel function in physically inactive adults. Isometric handgrip training is a promising strategy for lowering blood pressure and improving vascular health, but no previous investigations have studied the effect of training on markers of brain blood vessel function. Based on previous work showing improvements in vascular function after isometric handgrip training, we hypothesize that isometric handgrip training will improve key markers of cerebrovascular function.

DETAILED DESCRIPTION:
The incidence of cerebrovascular diseases is expected to increase. Early life sets the stage for vascular health outcomes later in life. Regular exercise is recommended for improving cerebrovascular health outcomes, but a lack of time or inadequate facilities are common exercise barriers. Not getting enough exercise is associated with worse cardiovascular and cerebrovascular health outcomes. There is a critical need for time-efficient strategies that require minimal equipment for improving cardiovascular and cerebrovascular health. Isometric handgrip (IHG) training is an effective strategy for improving cardiovascular health. Despite IHG's usefulness for improving vascular health through blood pressure reductions and improvements in endothelial function, almost nothing is known about IHG training and cerebrovascular function. Therefore, this project aims to test the hypothesis that 8 weeks of IHG training will improve cerebrovascular blood flow regulation and total cerebrovascular blood flow among adult humans who are not meeting the physical activity recommendations. We will measure middle cerebral artery blood velocity (MCAv) via transcranial Doppler ultrasound and assess MCAv dynamic autoregulation and MCAv reactivity to high and low carbon dioxide. We will also measure total cerebral blood flow, central artery stiffness, and MCAv pulsatility index. Understanding the effect of IHG on cerebrovascular health could inform exercise recommendations.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years old
* Body mass index ≤30 kg/m2 (without obesity)
* Physically inactive (not meeting the current recommendations of ≥150 minutes per week of moderate-to-vigorous aerobic exercise and not ≥2 days per week of resistance training) in last 6 months
* Have a smartphone and are willing to download mobile applications used in this project

Exclusion Criteria:

* Having an overt chronic condition (e.g., cardiovascular, cerebrovascular, etc.)
* Being pregnant, planning to become pregnant, or breastfeeding/lactating
* Regular use of nicotine products in the past 6 months
* Recent head injury/trauma or concussion

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-10-27 (Estimated); Study Completion 2028-10-27 (Estimated)

PRIMARY OUTCOMES:
Change in middle cerebral artery blood velocity reactivity to hypercapnia | Up to 9 weeks
  Middle cerebral artery blood velocity will be measured via transcranial Doppler ultrasound

SECONDARY OUTCOMES:
Change in middle cerebral artery blood velocity reactivity to hypocapnia | Up to 9 weeks
  Middle cerebral artery blood velocity will be measured via transcranial Doppler ultrasound
Brachial systolic blood pressure | Up to 9 weeks
  Blood pressure measured at the brachial artery
Change in dynamic cerebral autoregulation phase | Up to 9 weeks
  Calculated from middle cerebral artery blood velocity signal using transfer function analysis
Change in dynamic cerebral autoregulation gain | Up to 9 weeks
  Calculated from middle cerebral artery blood velocity signal using transfer function analysis
Change in total resting brain blood flow | Up to 9 weeks
  Total brain blood flow measured in the internal carotid and vertebral arteries at rest via ultrasound
Middle cerebral artery blood velocity pulsatility index | Up to 9 weeks
  Calculated from middle cerebral artery blood velocity signal

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided